CLINICAL TRIAL: NCT03775135
Title: Identity Development in Youth With Neuromuscular Diseases: A Clinically Relevant But Forgotten Issue in the Transition to Adulthood
Brief Title: Identity Development in Youth With Neuromuscular Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Changed plans
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S0000
Record Dates: First submitted 2018-11-13; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Neuromuscular Diseases
Keywords: Identity
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with neuromuscular diseases: Questionnaires will be administered by children with neuromuscular disease between 12 and 25 years and their parents
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Different questionnaires about identity development and psychosocial functioning will be administered

SUMMARY:
Up to 20% of the adolescents worldwide are diagnosed with a chronic illness. Although it's known that these young people suffer from a wide range of physical discomfort, in real life they have to cope with much more challenges whether or not caused by their physical situation. Psychiatric disorders (e.g. ASS, ADHD or depression) are more often diagnosed in this population compared to their healthy peers. The causal mechanisms for this higher risk, however, are yet unknown.

This project examines three underlying intrapersonal processes possibly having an impact on the evolution of these secondary symptoms. Previous research confirmed the significant impact of having a chronic illness on the development of identity and the association with a higher prevalence of depressive symptoms. Identity formation is a crucial developmental task to transfer from a child to an independent, responsible adult. We believe this developmental task is more at risk for youngsters and young adults suffering from a physical disability, caused by a neuromuscular disease. In this longitudinal research project, we investigate the development of identity in youth with a neuromuscular disease, compared to healthy peers and compared to a group of peers with a non-visible chronical illness. We also evaluate the impact of the degree of physical functioning on those mechanisms. Second, we examine if parental behavior and parental functioning is linked with the formation of identity in a neuromuscular populations. Finally, the impact of identity formation on psychosocial outcomes (e.g. feelings of depression and anxiety, quality of life, …) is measured.

By addressing these research questions, this project will add substantially to our knowledge on identity in chronic illness and can inform future prevention and intervention efforts targeting illness adaptation and parental functioning in order to prevent negative psychosocial outcomes and to optimize quality of life.

DETAILED DESCRIPTION:
A large-scale, multi-informant, two-wave longitudinal study is proposed to investigate our three different research objectives, using complementary methods and multiple sources for data collection. Such a longitudinal design allows for examining developmental trajectories of our core identity variables, as well as examining how these identity variables are related to other variables over time. As such, we will investigate integrative pathways linking contextual factors to identity development and broader psychosocial functioning, enabling us to forward important information for clinical practice. Before the start of the study, an approval from the ethical commission will be obtained. All data will be coded anonymously and stored in a confidential database. We aim to recruit 200 adolescents and emerging adults with a neuromuscular disease, like DMD patients (Duchenne Muscular Dystrophy), SMA patients (Spinal Muscular Atrophy), CMT patients (Charcot Marie Tooth) and MD1 patients (Myotonic Dystrophy, type 1). Patients will be included in this study if they meet the following criteria: confirmed diagnoses of a neuromuscular disorder; aged 12-25 years at baseline; last neuromuscular consult at our NMRC is 5 or less years ago; able to read and write Dutch; and valid contact details available in the clinical database or the hospital information system. Given the complex data-analyses, it is difficult to perform an exact power analysis, but the anticipated sample size is suited for the planned analyses (Kline, 2005). To make a useful comparison, we will include a control sample of age- and gender-matched healthy adolescents and a group of age- and gender-matched adolescents diagnosed with type 1 diabetes. Those control participants will be recruited in secondary schools and universities, while we are able to use the data of an ongoing research project in patients with diabetes. To achieve these aims, this project, as noted, will be in cooperation with the research team from the Faculty of Psychology and Educational Sciences at KU Leuven.

To investigate our objectives, data will be systematically collected during two years on two different occasions (T1 and T2), with one year between subsequent time-points. All neuromuscular patients are supposed to consult their multidisciplinary team every 6 months in the context of a general control and this gives us the opportunity to ask both adolescents and parents to complete questionnaires once a year. Depending on the date of the appointment, patients will start in this survey on different moments, but we will use the same time interval between time-points for every single patient. For inclusion, adolescents and parents will be asked to sign informed consents, where after demographic and clinical data can be obtained anonymously from the patients' medical records. Additional demographic and socio-economic information will be gathered using a demographic questionnaire at T1. Other data will be collected using instruments with well-established psychometric characteristics that mostly include self-reports on all two time-points (T1 and T2). Parents will also be asked to report on youth functioning as well. Figure 2 shows an overview of our research design and estimated timeline.

In order to investigate objective 1, adolescents will be asked to complete following questionnaires on the two different time-points: Dimensions of Identity Development Scale (25 items), Illness Identity Resolution Scale (27 items) and Brief Illness Perception Questionnaire (8 items). In addition, to examine reciprocal associations between identity development and the variables forwarded under objectives 2 en 3, adolescents will be asked to complete self-report questionnaires on psychosocial functioning and perceived support, using the Center for Epidemiologic Studies Depression Scale (CESD) (20 items) to screen for depressive symptoms, the Screen for Child Anxiety Related Emotional Disorders (SCARED-NL), the PedsQLTM Neuromuscular Module to measure quality of life and the Inventory of Peer and Parent Attachment: subscales Trust, Communication and Alienation (12 items). At the same time-points parents will be asked to complete the Illness Intrusive Scale (13 items), a scale about different factors of their parenting: responsiveness (7 items), psychological control (8 items), behavioral control (7 items) and overprotection/anxious parenting (8 items) (Parenting Questionnaire) and about the physical dependence of their child (Activ-Lim). To report about the psychosocial functioning of their child, parents will be asked to fulfill the Screen for Child Anxiety Related Emotional Disorders (SCARED-NL) and the PedsQLTM Neuromuscular Module to measure perceived quality of life in the youngster. For evaluating their own psychosocial functioning, they will be asked to complete the Center for Epidemiologic Studies Depression Scale (20 items) and a LAS-scale to evaluate their own quality of life. Necessary measures will be taken to minimize dropout: all participants receive a reward and Dillman's approach will be used to minimize non-response. Occasional missing data will be dealt with using appropriate methods (Enders, 2010). State-of-the-art longitudinal techniques will be used. Cross-lagged analysis will be used to examine directionality of effect, with appropriate controls for all within-time associations and stability coefficients. Hence, we can investigate, for instance, whether parents actually predict illness identity resolutions over time or whether reciprocal effects emerge with, for instance, illness acceptance also leading to more support. Further, mediation will be tested from a longitudinal perspective, allowing us to examine, for instance, whether illness identity resolutions mediate the associations between parental support and outcomes. To chart developmental trajectories over time, latent growth curve modeling estimates both linear and non-linear growth and uses information collected at all different time points to derive parameters of change (i.e., intercept and slope). Finally, latent class growth analysis will be used to identify distinct developmental trajectory classes in terms of personal and illness identity resolutions.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnoses of a neuromuscular disorder;
* aged 12-25 years at baseline;
* last neuromuscular consult at our NMRC is 5 or less years ago;
* able to read and write Dutch;
* valid contact details available in the clinical database or the hospital information system.

Exclusion criteria:

-Patients that do not fulfill the inclusion criteria

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with neuromuscular diseases between 12 and 25 years
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Manifestation of identity in 120 patients with neuromuscular diseases | up to year 1
  Identity development will be measured with specific questionnaires
Psychosocial functioning in 120 patients with neuromuscular diseases | up to year 1
  Psychosocial functioning will be measures with specific questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Goemans, MD, PhD, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: No